CLINICAL TRIAL: NCT00369161
Title: A Twelve-month, Multicenter, Open-label, Randomized Study of the Safety, Tolerability and Efficacy of Everolimus With IL-2 Receptor Antagonist, Corticosteroids and Two Different Exposure Levels of Tacrolimus in de Novo Renal Transplant Recipients
Brief Title: A Twelve-month, Multicenter, Open-label, Randomized Study of the Safety, Tolerability and Efficacy of Everolimus With Basiliximab, Corticosteroids and Two Different Exposure Levels of Tacrolimus in de Novo Renal Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRAD001A2426
Record Dates: First submitted 2006-08-25; First posted 2006-08-29 (Estimated); Results first posted 2011-01-19 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Renal Transplantation
MeSH Terms: interventions — Everolimus; Tacrolimus; Basiliximab; Adrenal Cortex Hormones

ARMS (2):
- Very low dose tacrolimus (Active Comparator): The first dose of everolimus was to be administered not later than 24 hours after transplantation with a starting dose of 1.5 mg bis in diem/twice a day (b.i.d.) thereafter adjusted to maintain the trough blood levels between 3 and 8 ng/ml. Tacrolimus was to be initiated within 24 hours after reperfusion of the graft with a starting dose of 0.1 mg/kg/day thereafter adjusted to maintain the trough blood levels between 4 and 7 ng/ml. Up to months three all patients received the same treatment and after three months patients in this arm received tacrolimus to reach a trough blood level between 1.5 and 3 ng/ml. All patients received two doses of 20 mg basiliximab, administered as an intravenous bolus injection. The first dose was given on the day of transplantation, with the second dose being administered on the fourth day post-transplant. Intravenous (i.v.) prednisone (or equivalent) was given pre- or intra-operatively according to center practice.
  Interventions: Drug: Everolimus (RAD001); Drug: Tacrolimus; Drug: Basiliximab; Drug: Corticosteroids
- Low dose tacrolimus (Active Comparator): The first dose of everolimus was to be administered not later than 24 hours after transplantation with a starting dose of 1.5 mg bis in diem/twice a day (b.i.d.) thereafter adjusted to maintain the trough blood levels between 3 and 8 ng/ml. Tacrolimus was to be initiated within 24 hours after reperfusion of the graft with a starting dose of 0.1 mg/kg/day thereafter adjusted to maintain the trough blood levels between 4 and 7 ng/ml. Up to months three all patients received the same treatment and after three months patients in this arm received tacrolimus to reach a trough blood level between 4 and 7 ng/ml. All patients received two doses of 20 mg basiliximab, administered as an intravenous bolus injection. The first dose was given on the day of transplantation, with the second dose being administered on the fourth day post-transplant. Intravenous (i.v.) prednisone (or equivalent) was given pre- or intra-operatively according to center practice.
  Interventions: Drug: Everolimus (RAD001); Drug: Tacrolimus; Drug: Basiliximab; Drug: Corticosteroids

INTERVENTIONS:
Drug: Everolimus (RAD001)
Drug: Tacrolimus
Drug: Basiliximab
Drug: Corticosteroids

SUMMARY:
This study is designed to evaluate whether tacrolimus dose reduction in de novo renal recipients receiving everolimus can preserve renal function while maintaining efficacy.

ELIGIBILITY:
Inclusion criteria

* Male or female of 18-65 years old
* Patient who has received a primary kidney transplant from a cadaveric, living unrelated or non-human leucocyte antigen (HLA) identical living related donor
* Recipient of a kidney with a cold ischemia time (CIT) < 30 hours
* Recipient of a kidney from a donor 10-65 years old
* Patient able to receive the first dose of tacrolimus within 24 hours from graft reperfusion
* Female capable of becoming pregnant must have a negative pregnancy test and is required to practice a medically approved method of birth control for the duration of the study and for a period of three months following discontinuation of investigational drug
* Patient willing and capable of giving written informed consent for study participation and able to participate in the study for 12 months

Exclusion criteria

* Patient who has previously received an organ transplant
* Recipient of multiple organ transplants
* Recipient of a kidney transplant from a non heart-beating donor
* Recipient of donor specific transfusions
* Recipient of A-B-O incompatible transplant or T-cell cross-match positive transplant
* Patient with current Panel Reactive Antibodies (PRA) level ≥ 50%
* Recipient of a kidney from a donor who tests positive for hepatitis B surface antigen or hepatitis C antibodies
* Patient who is human immunodeficiency virus (HIV) positive
* Patient who has a positive hepatitis C serology or who is hepatitis B surface antigen positive with evidence of liver injury as indicated by aspartate aminotransferase (AST)/alanine aminotransferase (ALT) levels ≥2.5 times upper limit of normal (UNL). Viral serology results obtained within 6 months prior to the administration of the first dose of Certican™ are acceptable
* Patient with severe hypercholesterolemia (350 mg/dL, 9.1 mmoL/dL) or hypertriglyceridemia ( 500 mg/dL, 5.6 mmoL/L)
* Patient with white blood cell (WBC) count 3,000/mm3 or with platelet count 75,000/mm3
* Patient with any severe allergy requiring acute (within 4 weeks of baseline) or chronic treatment, or with hypersensitivity to drugs similar to Certican (e.g., macrolides)
* Patient who has been treated with an immunosuppressive drug or an investigational drug within 4 weeks prior to the administration of the first dose of Certican
* Patient with uncontrolled infection
* Patient with any surgical or medical condition, other than the current transplant, which in the opinion of the investigator, precludes enrollment in this trial
* Patient with a known malignancy or a history of malignancy within last 5 years other than successfully treated localized basal or squamous cell carcinoma of the skin
* Abnormal physical or laboratory findings of clinical significance within 2 weeks prior to the administration of the first dose of Certican™ which at investigator's discretion would interfere with the objectives of the study
* Breast feeding women
* Patient with symptoms of significant somatic or mental illness or with unresolved history of drug or alcohol abuse
* Patient unable to cooperate or communicate with the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2006-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis, Basel, Switzerland

REFERENCES:
- [Derived] Langer RM, Hene R, Vitko S, Christiaans M, Tedesco-Silva H Jr, Ciechanowski K, Cassuto E, Rostaing L, Vilatoba M, Machein U, Ulbricht B, Junge G, Dong G, Pascual J. Everolimus plus early tacrolimus minimization: a phase III, randomized, open-label, multicentre trial in renal transplantation. Transpl Int. 2012 May;25(5):592-602. doi: 10.1111/j.1432-2277.2012.01465.x. Epub 2012 Mar 26. PMID 22471345

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Centers in 13 countries screened at least 1 patient: Argentina, Brazil, Chile, Czech Republic, France, Hungary, Mexico, The Netherlands, Poland, Portugal, South Africa, Spain,Turkey. Starting 27 June 2006 and ending 29 Dec 2008.
Groups:
- Low Dose Tacrolimus: The first dose of everolimus was to be administered not later than 24 hours after transplantation with a starting dose of 1.5 mg bis in diem/twice a day (b.i.d) thereafter adjusted to maintain the trough blood levels between 3 and 8 ng/ml. Tacrolimus was to be initiated within 24 hours after reperfusion of the graft with a starting dose of 0.1 mg/kg/day thereafter adjusted to maintain the trough blood levels between 4 and 7 ng/ml. Up to months three all patients received the same treatment and after three months patients in this arm received tacrolimus to reach a trough blood level between 4 and 7 ng/ml. All patients received two doses of 20 mg basiliximab, administered as an intravenous bolus injection. The first dose was given on the day of transplantation, with the second dose being administered on the fourth day post-transplant. Intravenous (i.v.) prednisone (or equivalent) was given pre- or intra-operatively according to center practice.
Period: Overall Study
Arm/Group | Very Low Dose Tacrolimus | Low Dose Tacrolimus
Started | 109 ("Started" indicates randomized and safety population.) | 119
Intention to Treat (ITT) | 107 | 117
Completed | 82 | 95
Not Completed | 27 | 24
Not completed — Adverse Event | 15 | 13
Not completed — Abnormal laboratory value | 0 | 1
Not completed — Lack of Efficacy | 3 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Death | 1 | 2
Not completed — Graft loss | 4 | 0
Not completed — Administrative Problem | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Very Low Dose Tacrolimus | Low Dose Tacrolimus | Total
Number analyzed (Participants) | 107 | 117 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] — Baseline measures are based on intention to treat (ITT) population.
  years | 44.6 (12.75) | 46.9 (12.08) | 45.8 (12.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 48 | 96
  Male | 59 | 69 | 128

OUTCOME MEASURES:

1. Primary Outcome: Renal Function Assessed by Calculated Glomerular Filtration Rate (cGFR)
Description: Renal function was assessed by calculated glomerular filtration rate (cGFR) using Modification of Diet in Renal Disease (MDRD)formula.
  GFR [mL/min/1.73m^2] = 186.3*(C-1.154)*(A-0.203)*G*R, where:
  * C is the serum concentration of creatinine [mg/dL],
  * A is patient age at sample collection date [years],
  * G=0.742 when gender is female, otherwise G=1,
  * R=1.21 when race is black, otherwise R=1
Time Frame: 12 months post -transplant
Population: Modified Intent-to-treat (ITT) population i.e patients with an available cGFR at month 12.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Very Low Dose Tacrolimus | Low Dose Tacrolimus
Number analyzed (Participants) | 92 | 105
mL/min/1.73m^2 | 57.07 (19.467) | 51.73 (19.995)

2. Secondary Outcome: Number of Participants With Incidence of Biopsy-proven Acute Rejection (BPAR)
Description: Biopsy-proven acute rejection (BPAR) was defined as a clinically suspected acute rejection confirmed by biopsy (performed by the local pathologist). For all clinically suspected rejection episodes a graft core biopsy must have been performed before or within a 24 hour period from the initiation of anti-rejection therapy.
Time Frame: from Month 4 through to Month 12
Population: Intention to treat (ITT) population.
Measure: Number; unit: participants
Arm/Group | Very Low Dose Tacrolimus | Low Dose Tacrolimus
Number analyzed (Participants) | 107 | 117
participants | 2 | 1

3. Secondary Outcome: Percentage of Participants With Efficacy Failure
Description: Efficacy failure was a composite of BPAR, graft loss, death or lost to follow-up. BPAR was defined as a clinically suspected acute rejection confirmed by biopsy (performed by the local pathologist). For all clinically suspected rejection episodes a graft core biopsy must have been performed before or within a 24 hour period from the initiation of anti-rejection therapy. An allograft was presumed to be lost on the day a patient started dialysis and was unable to subsequently be removed from dialysis. If the patient underwent a graft nephrectomy, the day of nephrectomy was the day of graft loss.
Time Frame: Month 12
Population: Intention to treat (ITT) population.
Measure: Number; unit: percentage of participants
Arm/Group | Very Low Dose Tacrolimus | Low Dose Tacrolimus
Number analyzed (Participants) | 107 | 117
percentage of participants
  Efficacy failure (Composite) | 6.7 | 4.3
  BPAR | 2.7 | 1.1
  Graft loss or death | 4.0 | 2.2
  Graft Loss | 1.3 | 1.1
  Death | 2.7 | 1.1
  Lost To Follow-up | 0.0 | 1.1

ADVERSE EVENTS:
Description: All randomized patients who are also considered as safety population
Arm/Group | Very Low Dose Tacrolimus | Low Dose Tacrolimus
Serious Adverse Events (participants affected / at risk) | 64/109 | 61/119
Other Adverse Events (participants affected / at risk) | 103/109 | 114/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Very Low Dose Tacrolimus (N=109) | Low Dose Tacrolimus (N=119)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Haemolysis (Blood and lymphatic system disorders) | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 | 2
Lymphatic disorder (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Giant cell epulis (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 2
Pyrexia (General disorders) | 3 | 4
Kidney transplant rejection (Immune system disorders) | 2 | 0
Transplant rejection (Immune system disorders) | 2 | 0
Abscess intestinal (Infections and infestations) | 1 | 0
Acute tonsillitis (Infections and infestations) | 1 | 0
Arteriovenous graft site infection (Infections and infestations) | 1 | 0
BK virus infection (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 1 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 2 | 2
Encephalitis viral (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Hepatitis E (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 2
Infected lymphocele (Infections and infestations) | 0 | 2
Lung infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 4
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0
Postoperative abscess (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 2 | 4
Septic shock (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Superinfection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 10 | 13
Urosepsis (Infections and infestations) | 2 | 2
Wound infection (Infections and infestations) | 1 | 2
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 8 | 7
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 1
Graft complication (Injury, poisoning and procedural complications) | 1 | 1
Graft loss (Injury, poisoning and procedural complications) | 0 | 1
Graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 7 | 13
Cytomegalovirus test (Investigations) | 0 | 1
Renal function test abnormal (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Weight increased (Investigations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 4 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 2
Ischaemic stroke (Nervous system disorders) | 0 | 1
Paraplegia (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Acute psychosis (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Anuria (Renal and urinary disorders) | 0 | 1
Bladder stenosis (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 1
Nephropathy (Renal and urinary disorders) | 0 | 1
Obstructive uropathy (Renal and urinary disorders) | 1 | 1
Reflux nephropathy (Renal and urinary disorders) | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 1 | 0
Renal artery thrombosis (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 2
Renal tubular disorder (Renal and urinary disorders) | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0
Ureteral necrosis (Renal and urinary disorders) | 1 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 1
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary vasculitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 2 | 0
Iliac artery stenosis (Vascular disorders) | 1 | 1
Ischaemia (Vascular disorders) | 1 | 0
Lymphocele (Vascular disorders) | 2 | 6
Phlebitis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 1
Vasculitis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Very Low Dose Tacrolimus (N=109) | Low Dose Tacrolimus (N=119)
Anaemia (Blood and lymphatic system disorders) | 29 | 28
Abdominal pain (Gastrointestinal disorders) | 7 | 7
Abdominal pain upper (Gastrointestinal disorders) | 2 | 6
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 7
Constipation (Gastrointestinal disorders) | 15 | 22
Diarrhoea (Gastrointestinal disorders) | 17 | 19
Nausea (Gastrointestinal disorders) | 7 | 7
Vomiting (Gastrointestinal disorders) | 7 | 2
Oedema (General disorders) | 9 | 13
Oedema peripheral (General disorders) | 25 | 27
Pyrexia (General disorders) | 11 | 17
Nasopharyngitis (Infections and infestations) | 7 | 4
Upper respiratory tract infection (Infections and infestations) | 1 | 9
Urinary tract infection (Infections and infestations) | 29 | 34
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 15 | 11
Graft complication (Injury, poisoning and procedural complications) | 7 | 4
Post procedural haematoma (Injury, poisoning and procedural complications) | 7 | 4
Procedural pain (Injury, poisoning and procedural complications) | 12 | 12
Wound complication (Injury, poisoning and procedural complications) | 5 | 6
Blood creatinine increased (Investigations) | 5 | 9
Acidosis (Metabolism and nutrition disorders) | 6 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 10 | 16
Dyslipidaemia (Metabolism and nutrition disorders) | 14 | 21
Hypercholesterolaemia (Metabolism and nutrition disorders) | 23 | 31
Hyperglycaemia (Metabolism and nutrition disorders) | 15 | 13
Hyperkalaemia (Metabolism and nutrition disorders) | 14 | 11
Hyperlipidaemia (Metabolism and nutrition disorders) | 15 | 19
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 6 | 15
Hyperuricaemia (Metabolism and nutrition disorders) | 6 | 11
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 17 | 16
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 7
Iron deficiency (Metabolism and nutrition disorders) | 3 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 7
Osteoporosis (Musculoskeletal and connective tissue disorders) | 6 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 6
Headache (Nervous system disorders) | 11 | 9
Tremor (Nervous system disorders) | 6 | 3
Insomnia (Psychiatric disorders) | 12 | 20
Dysuria (Renal and urinary disorders) | 6 | 8
Proteinuria (Renal and urinary disorders) | 12 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Acne (Skin and subcutaneous tissue disorders) | 15 | 6
Hypertension (Vascular disorders) | 17 | 19
Lymphocele (Vascular disorders) | 7 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial; or publication of the trial results in their entirety.